CLINICAL TRIAL: NCT04948177
Title: Outcome of Gastric Fundus and Pylorus Botulinum Toxin A Injection in Obese Patients Class I-II With Normal Pyloric Orifice Structure: A Retrospective Analysis
Brief Title: Outcome of Gastric Fundus and Pylorus Botulinum Toxin A Injection
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, M.D, Asisstant Professor, Assistant Director of Transplantation Clinic, Okan University
Other Study IDs: 56665618-204.01.07A
Record Dates: First submitted 2021-06-19; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Group A: Individuals who had normal pyloric orifice structure;
- Group B: Group B: Individuals who have abnormal pyloric orifice structure

SUMMARY:
Newly, botulinum toxin A application into the stomach has been proposed as a treatment method in obesity. It impacts through acetylcholine receptors located in smooth muscle cells and suppresses stomach motility. This method aims to decrease gastric emptying time and thus to extend the duration of feeling full. This effect of intragastric botulinum toxin A injection (GBI) makes it easier to adhere to dietary prescriptions, which is the cornerstone of any obesity treatment method.

Endoscopic inspections and the complicatedness in literature results, cases that have not succeeded in losing weight after GBI might have pylorus contractility problems. Any deterioration in pylorus activity is recognized to have the potential to influence gastric emptying. In such a case, gastric emptying time would also be altered due to the paralysis of pylorus muscles, which is one of the effect mechanisms of botulinum toxin A.

The pyloric orifice structure may have a crucial role in the success or failure of GBI therapy for obesity treatment.

DETAILED DESCRIPTION:
The prevalence of obesity has doubled globally in the last four decades to the extent that nearly one-third of the world population is now classified as overweight/obese. Obesity causes adverse impacts on almost every physiological system in the human body and comprises an important public health problem. It is associated with an increased risk of many developing co-morbid conditions, such as diabetes mellitus, cardiovascular disease, several types of cancers, musculoskeletal disorders, and poor mental health.

Current treatment options for patients with obesity include lifestyle intervention, obesity pharmacotherapy, and bariatric surgery. The components of lifestyle intervention involve diet, exercise, and behavior modification and should be recognized as the cornerstone of any obesity treatment method; however, the impact of lifestyle intervention is limited in patients with morbid obesity.

Surgical therapies with laparoscopic approach are accepted as the most effective and persistent obesity-treatment methods, with a significant reduction in complication rates and postoperative recovery. Gastric banding, sleeve gastrectomy, Roux-en-Y gastric bypass, and biliopancreatic diversion are commonly performed bariatric surgical procedures worldwide. But, the idea of scarless methods in which the video-endoscopy device is used as the primary carrier device, expecting to achieve results at least as good as laparoscopic procedures, has significantly developed within the last decade. Additionally, the development of effective and safe, newer endoscopic bariatric procedures provides another adjunctive treatment for patients with obesity who cannot handle this disease with lifestyle modification alone or who is not a candidate for surgical procedures. Endoscopic therapies, such as intra-gastric balloons, duodenojejunal bypass liners such as the EndoBarrier, and endoscopic suturing platforms, have also become proposed alternatives to surgery, considering their minimally-invasive advantages. However, given the lack of long-term data at present, the role of such devices continues to be determined.

Newly, botulinum toxin A application into the stomach has been proposed as a treatment method in obesity. It impacts through acetylcholine receptors located in smooth muscle cells and suppresses stomach motility. This method aims to decrease gastric emptying time and thus to extend the duration of feeling full. This effect of intragastric botulinum toxin A injection (GBI) makes it easier to adhere to dietary prescriptions, which is the cornerstone of any obesity treatment method.

Endoscopic inspections and the complicatedness in literature results, cases that have not succeeded in losing weight after GBI might have pylorus contractility problems. Any deterioration in pylorus activity is recognized to have the potential to influence gastric emptying. In such a case, gastric emptying time would also be altered due to the paralysis of pylorus muscles, which is one of the effect mechanisms of botulinum toxin A.

The pyloric orifice structure may have a crucial role in the success or failure of GBI therapy for obesity treatment.

The present study aims to explore whether there is a correlation between weight loss after GBI and pyloric orifice structure.

ELIGIBILITY:
Inclusion Criteria:

-Class I obese patients and class II obese patients with no comorbidities

Exclusion Criteria:

* Patients with type 3-4 hiatal hernia according to flap-valve grading system
* Los Angeles type B-C esophagitis
* Type I-II ulcer
* Malignant or suspected malignant lesion in stomach
* Age <18 or >70
* Patients use drugs affecting gastric contractility and pyrokinesis
* Patients have endocrine system problems (hypothyroidism and Cushing syndrome), active psychiatric disorder were not accepted as a candidate for GBI therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records of patients who underwent intragastric botulinum toxin A from June 2019 through June 2020 at the Okan University Hospital in Istanbul were retrospectively evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index Change | 6 months
  The body mass index change in six months period is observed

SECONDARY OUTCOMES:
Weight change | 6 months
  The weight change in six months period is observed

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)